CLINICAL TRIAL: NCT03487146
Title: Hemoperfusion in Combination With Hemodialysis for Improvement of Self-reported Sleep Disturbance and Overall Survival Rate in Maintenance Hemodialysis Patients
Brief Title: HP Improves Sleep and Overall Survival Rate in Maintenance Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Principal Investigator, Jin HM, MD, Professor, Shanghai Pudong Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiPudongH1
Record Dates: First submitted 2018-03-26; First posted 2018-04-03 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Hemoperfusion
MeSH Terms: interventions — Hemoperfusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HD(hemodialysis) group (No Intervention): HD group as conventional control arm
- HD+HP(hemodialysis+hemoperfusion) group (Active Comparator): HD+HP as active interventional group.HP was performed 1-2 times/per 2 weeks, and each session lasted for two hours.
  Interventions: Device: hemoperfusion(HP)

INTERVENTIONS:
Device: hemoperfusion(HP) — These patients were computer-matched into two groups, involving 100 patients with absolute HD vs. 100 cases with HD+HP.HP was performed 1-2 times/per 2 weeks, and each session lasted for two hours.Self-reported sleep disturbance was evaluated before and after observational time (two-year period), which lasted at least 7 hours based on the recommendations presented by National Institute of Health (NIH). Sleep efficiency (%) was calculated as the ratio of sleep duration to total time in bed, and was multiplied by 100.
  Arms: HD+HP(hemodialysis+hemoperfusion) group

SUMMARY:
Sleep disturbance has been long-standing torments in most of patients with maintenance hemodialysis (HD). In this study, we attempted to explore whether long-term hemoperfusion (HP) could improve sleep disorder and increase overall survival rate in HD patients.

ELIGIBILITY:
Inclusion Criteria:

1. duration of maintenance HD should be equal or more than 3 months,
2. patient's age should be equal or more than 18 years

   Exclusion Criteria:

   - i) he/she diagnosed with malignant tumors, an active rheumatism, infectious diseases, or a severe heart failure ii) he/she would disagree with the study
3. he/she has received a short-term poor prognosis
4. he/she would be more than 80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
improvement of self-reported sleep disturbance | 2 years
  Analysis of the sleep disturbance by using Pittsburgh Sleep Quality Index (PSQI) questionnaire

SECONDARY OUTCOMES:
survival | 2 years
  increase overall survival rate